CLINICAL TRIAL: NCT05324267
Title: Analysis of the Determinants of Sleep Quality in a Spanish Population. a Study Protocol for a Cross-sectional Study
Brief Title: Determinants of Sleep Quality in Spanish Population (SSQD Study)
Acronym: SSQD
Status: Completed | Type: Observational
Sponsor: University of Salamanca (Other)
Collaborators: Gerencia Regional de Salud de Castilla y Leon (Other); Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Principal Investigator, José Ignacio Recio Rodriguez, PhD, Associate Professor, University of Salamanca
Other Study IDs: GRS 2320/A/21
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Sleep Quality
Keywords: Life Style; Psychological Factors; Melatonin
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Introduction: Sleep disorders are a growing concern for public health, being related, among others, to an increased risk of cardiovascular diseases or poorer cognitive functioning. In addition, these might have a possible impact on aspects related to personal motivation and quality of life. However, few studies have analyzed the possible determinants of sleep quality in the adult population as a whole, establishing patterns based on these.

Objective: To evaluate the determinants of sleep quality in a representative sample of the general adult population aged 25 to 65 years old and to establish patterns of sleep quality based on lifestyles, psychological factors, morbidities and biological markers.

Methodology:

Design: This is a descriptive observational, cross-sectional study that will include a representative sample of 500 people aged 25 to 65 years old from the city of Salamanca (Spain) selected by random sampling stratified by age and sex.

Study variables: A visit lasting approximately 90 minutes will be carried out. The determinants of sleep quality will be assessed using both objective and self-reported methods. Variables related to life styles will be assessed: physical activity, diet and toxic habits including tobacco smoking or alcohol use. Morbidity data will also be collected, and psychological factors such as anxiety will also be assessed. Serum melatonin levels will be determined as a biological marker related to sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-65 years old
* Sign the informed consent

Exclusion Criteria:

* Patients with terminal disease
* Any clinical condition that would interfere with study procedures

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include participants affiliated with the Health Service of Castilla y León (SACYL) (Spain) who meet all the eligibility criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Sleep quality | Baseline
  Measured by accelerometer (Actigraph GT3X). This device reports Total Sleep Time (TST) measured in minutes.
Sleep quality | Baseline
  Measured by the Pittsburgh Sleep Quality Index (PSQI). Possible scores on the PSQI range from 0 (no difficulty) to 21 (severe difficulties in all areas).

SECONDARY OUTCOMES:
Physical activity | Baseline
  Measured by accelerometer (Actigraph GT3X). This device reports physical activity measured in steps per hour.
Diet | Baseline
  Measured by the Mediterranean Diet Adherence Screener (MEDAS). Possible scores range from 0 (lower adherence) to 14 (higher adherence).
Tobacco smoking | Baseline
  Measured by the Fagerström Test for Nicotine Dependence. This six-item questionnaire generates test scores ranging from 0 to 10, with higher scores indicating greater nicotine dependence.
Alcohol use | Baseline
  Measured by the Alcohol Use Disorders Identification Test (AUDIT). Possible scores range from 0 to 40. An AUDIT score of 8 or more indicates hazardous or harmful alcohol use; a score of less than 8 indicates non-hazardous consumption.
Anxiety | Baseline
  Measured by the Generalized Anxiety Disorder (GAD-7) questionnaire. Possible scores range from 0 to 21. Increasing scores indicate higher levels of anxiety.
Serum melatonin levels | Baseline
  Serum melatonin levels (measured in pg/ml) will be determined by high performance liquid chromatography-triple quadrupole mass spectrometry (HPLC-MS/MS triple quadrupole).

CONTACTS AND LOCATIONS:
Locations (1):
- José Ignacio Recio Rodriguez, Salamanca, Salamanca, Spain

REFERENCES:
- [Derived] Jimenez-Vaquero C, Gonzalez-Sanchez J, Alonso-Dominguez R, Garcia-Yu IA, Sanchez-Aguadero N, Crespo-Sedano A, Rihuete-Galve MI, Recio-Rodriguez JI. Sleep quality in Spanish adults: an age- and sex-stratified cross-sectional study. Sci Rep. 2025 Dec 12;15(1):43670. doi: 10.1038/s41598-025-27418-7. PMID 41387971
- [Derived] Jimenez-Vaquero C, Gonzalez-Sanchez J, Alonso-Dominguez R, Garcia-Yu IA, Sanchez-Aguadero N, Crespo-Sedano A, Rihuete-Galve MI, Recio-Rodriguez JI. Sex-specific sleep profiles in Spanish adults: cross-sectional actigraphy-PSQI study with cluster analysis in Salamanca and Avila. BMJ Open. 2025 Nov 4;15(11):e103094. doi: 10.1136/bmjopen-2025-103094. PMID 41248358
- [Derived] Jimenez-Vaquero C, Alonso-Dominguez R, Garcia-Yu IA, Martin-Nogueras AM, Sanchez-Aguadero N, Crespo-Sedano A, Rihuete-Galve MI, Garcia-Alonso MA, Garcia-Prieto ML, Gonzalez-Sanchez J, Recio JI. Analysis of the determinants of sleep quality in a Spanish population: a study protocol for a cross-sectional study. BMJ Open. 2023 Mar 8;13(3):e069444. doi: 10.1136/bmjopen-2022-069444. PMID 36889827